CLINICAL TRIAL: NCT00073489
Title: A Pilot Trial of OSI-461 in Patients With Chronic Lymphocytic Leukemia
Brief Title: A Pilot Study of OSI-461 in Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-005; NCT00036049 (obsolete NCT alias)
Record Dates: First submitted 2003-11-21; First posted 2003-11-25 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic leukemia; leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: OSI-461

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of OSI-461 in CLL patients.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the activity of OSI-461 given twice daily orally in previously untreated CLL patients. The secondary objective is to evaluate the safety profile of OSI-461 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL established by bone marrow aspiration and biopsy or flow cytometry of peripheral blood.
* No previous therapy for CLL.
* Expected remaining life span greater than or equal to six months.
* 18 years or older.
* Willingness and ability to sign an informed consent.

Exclusion Criteria:

* Other active malignancy or history of treatment of any malignancy (excluding non-melanoma skin cancer) within the previous three years.
* History of other malignancy which could affect the diagnosis or assessment of OSI-461.
* Previous therapy for CLL.
* Use of an investigational medication or device within one month of initiating study therapy.
* Concurrent immunotherapy.
* Use of steroids at the time of enrollment (patients who require steroids after enrollment may remain on study).
* Any condition or any medication which may interfere with the conduct of the study.
* Serious uncontrolled intercurrent medical or psychiatric illness, including serious infection.
* Evidence of CNS involvement.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23
Dates: Start 2001-05; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Arizona Hematology & Oncology Associates, Phoenix, Arizona
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Florida Oncology Associates, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Iowa Oncology Associates, Cedar Rapids, Iowa
  - Oncology/Hematology Associates of Kansas City, Kansas City, Missouri
  - Piedmont Hem Onc Assoc, P.A., Winston-Salem, North Carolina
  - Dayton Oncology/Hematology Consultants, Dayton, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Southwest Regional Cancer Center, Austin, Texas
  - Hematology Oncology Associates of South Texas, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Cancer Care Northwest, Spokane, Washington